## INTERNATIONAL REGISTRY FOR AMBULATORY BLOOD PRESSURE AND ARTERIAL STIFFNESS TELEMONITORING (VASOTENS REGISTRY)

| Patient number: | Initials: | Date: | 1 | / | |
|-----------------|-----------|-------|-----|-------|------|
| | | | DAY | MONTH | YEAR |

## INFORMED CONSENT FORM version 1.0 28/01/2015

## **Declaration of consent**

I have read the foregoing information, or it has been read to me. I declare that I have understood all the information relating to the present clinical research, and that I have had the opportunity to ask questions about it and any questions that I have asked have been answered to my satisfaction.

I consent voluntarily to participate in the study, knowing that such participation is voluntary and that I can withdraw at any time.

I agree to provide laboratory examinations and blood tests performed before entering the study.

By signing this form I agree also to handle my personal data for research purposes to the extent and in the manner indicated in the information sheet provided to me with the present document.

I will receive a copy of the present informed consent form, after signing.

PARTICIPANT'S SURNAME AND NAME

(in block letters)

SIGNATURE

DATE

(day/month/year)

I have accurately read out the information sheet to the potential participant, and to the best of my ability made sure that the participant understood the procedures of the study. I confirm that the participant was given an opportunity to ask questions about the study, and all the questions asked by the participant have been answered correctly and to the best of my ability. I confirm that the individual has not been coerced into giving consent, and the consent has been given freely and voluntarily.

A copy of this Informed Consent Form has been provided to the participant.

INVESTIGATOR'S SURNAME AND NAME

(in block letters)

INVESTIGATOR'S SIGNATURE

DATE

(day/month/year)